CLINICAL TRIAL: NCT01149096
Title: A Comparison of Acute and Long-term Toxicities in Bone Marrow Donors With and Without G-CSF Treatment Prior to Harvest: A Companion Study to ASCT0631
Brief Title: Collection of Bone Marrow From Donors Treated With or Without Filgrastim
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ASCT0631D; NCI-2011-02237 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000675536; COG-ASCT0631D; ASCT0631D (Other: Childrens Oncology Group); ASCT0631D (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2019-09

CONDITIONS: Healthy Stem Cell Donor; No Evidence of Disease
MeSH Terms: interventions — Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (conventional bone marrow harvest) (Active Comparator): Donors undergo conventional (i.e., unstimulated) bone marrow harvest on day 0.
  Interventions: Procedure: Bone Marrow Donation; Other: Laboratory Biomarker Analysis
- Arm II (filgrastim, bone marrow harvest) (Experimental): Donors receive filgrastim subcutaneously on days -4 through 0. Donors then undergo bone marrow harvest on day 0.
  Interventions: Procedure: Bone Marrow Donation; Biological: Filgrastim; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Bone Marrow Donation — Undergo bone marrow harvest
Biological: Filgrastim — Given subcutaneously
  Other Names: G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
  Arms: Arm II (filgrastim, bone marrow harvest)
Other: Laboratory Biomarker Analysis — Optional correlative studies

SUMMARY:
This randomized clinical trial is studying the side effects of collection of bone marrow from donors treated with or without filgrastim. Giving colony-stimulating factors, such as filgrastim (G-CSF), to donors helps the stem cells move from the bone marrow to the blood so they can be collected and stored.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate short- and long-term toxicities in bone marrow donors treated with vs without filgrastim before harvest.

II. To compare 10-year mortality and cancer in donors treated with vs without filgrastim.

SECONDARY OBJECTIVES:

I. To correlate the incidence of acute and chronic graft-vs-host disease in the marrow recipients enrolled on COG-ASCT0631 with four parameters assessed in the bone marrow harvests: absolute T-cell numbers, Th1 vs Th2 profile of T-cells, dendritic cell populations, and T-regulatory cell content.

OUTLINE: Donors are randomized to 1 of 2 treatment arms.

ARM I (unstimulated harvest): Donors undergo conventional (i.e., unstimulated) bone marrow harvest on day 0.

ARM II (stimulated harvest): Donors receive filgrastim subcutaneously on days -4 through 0. Donors then undergo bone marrow harvest on day 0.

After completion of study treatment, donors are followed up at 1, 6, and 12 months and then annually for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Appropriately human leukocyte antigen (HLA)-matched (HLA, A, B, DRB1 identical or antigen mismatched [i.e., 5/6 or 6/6 antigens matched]) sibling of the bone marrow recipient enrolled on COG-ASCT0631
* Adequate size relative to the recipient (i.e., harvesting the maximum of 20 cc/kg from the donor would result in a bone marrow graft that will provide an adequate cell and volume dose to the recipient, in the opinion of the treating physician)
* Enrolled on the COG Umbrella Long-Term Follow-Up Study COG-ALTE05N1
* Not pregnant or nursing
* No human immunodeficiency virus (HIV) positivity
* No sickle cell trait or sickle cell anemia/disease
* Not at an increased risk from bone marrow donation after filgrastim administration due to a pre-existing medical condition, as determined by an independent physician separate from the research team
* None of the following:

  * Active infection, especially pulmonary
  * Splenomegaly or a history of splenic injury
  * Active or recent pulmonary disease (i.e., pneumonia within the past 4 weeks)
  * A condition that would make the donor unsuitable to donate, as determined by an independent physician separate from the research team
* No autoimmune disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-06-14 (Actual); Primary Completion 2011-12-14 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan A Grupp, Principal Investigator — Children's Oncology Group
Locations (22):
- United States (22):
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Norton Children's Hospital, Louisville, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Childrens Oncology Group, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Primary Children's Hospital, Salt Lake City, Utah
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Conventional Bone Marrow Harvest) | Arm II (Filgrastim, Bone Marrow Harvest)
Started | 6 | 7
Completed | 6 | 6
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Conventional Bone Marrow Harvest) | Arm II (Filgrastim, Bone Marrow Harvest) | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 5 | 11
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.5 (5.2) | 14.4 (5.9) | 10.8 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Short-term Adverse Events in G-CSF (Filgrastim) Stimulated Bone Marrow (G-BM) Donors
Description: The Kaplan-Meier method will be used to estimate the cumulative incidence of short term adverse events defined by having any of the following events: 1) death due to a cause that is unknown or possibly related to G-CSF, 2) development of a malignancy, 3) development of a splenic rupture, or 4) development of a severe acute lung injury possibly related to GCSF therapy.
Time Frame: Up to 1 year after donation
Population: Analysis conducted within G-BM donors only, therefore, no report for the control arm (Conventional bone marrow transplant).
Measure: Number; unit: Percentage of patients
Arm/Group | Arm II (Filgrastim, Bone Marrow Harvest)
Number analyzed (Participants) | 7
Percentage of patients | 0

2. Primary Outcome: Percentage of Participants Who Experienced Death in G-CSF Stimulated-bone Marrow (G-BM) Donors
Description: The Kaplan-Meier method will be used to estimate the cumulative incidence of death event in G-BM donors only.
Time Frame: Up to 1 year after donation
Population: Analysis conducted for stimulated-bone marrow (G-BM) donors only, therefore, no report on the control arm (Conventional bone marrow transplant).
Measure: Number; unit: Percentage of patients
Arm/Group | Arm II (Filgrastim, Bone Marrow Harvest)
Number analyzed (Participants) | 7
Percentage of patients | 0

3. Primary Outcome: Percentage of Participants With Grade 1 or 2 Toxicities
Description: Estimate the percentage of patients having non-fatal complications of CTCAE Grades 1 or 2 in standard BM and G-CSF stimulated-bone marrow (G-BM) donors.
Time Frame: Up to 1 year after donation
Population: Modified Toxicity Criteria and Pain Assessment was used with higher grades corresponding to more severe AEs.
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (Conventional Bone Marrow Harvest) | Arm II (Filgrastim, Bone Marrow Harvest)
Number analyzed (Participants) | 6 | 7
percentage of patients | 67 | 86

4. Primary Outcome: Percentage of Participants With Grade 3 or 4 Toxicities
Description: Estimate the percentage of patients having non-fatal complications of Grade 3 other than pain (consider Grade 4 for pain only), or any of Grade 4 in standard BM and G-CSF stimulated-bone marrow (G-BM) donors. Modified Toxicity Criteria and Pain Assessment was used with higher grades corresponding to more severe AEs.
Time Frame: Up to 1 year after donation
Population: All patients included in analysis. No incidence of grades 3 or 4 toxicities.
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (Conventional Bone Marrow Harvest) | Arm II (Filgrastim, Bone Marrow Harvest)
Number analyzed (Participants) | 6 | 7
percentage of patients | 0 | 0

5. Primary Outcome: 10-year Mortality Rate in Marrow Donors
Description: The Kaplan-Meier method will be used to estimate overall survival probabilities in standard BM and G-BM donors.
Time Frame: Up to 10 years post bone marrow harvest
Population: Data were not collected as no patients were followed to 10 years.
Arm/Group | Arm I (Conventional Bone Marrow Harvest) | Arm II (Filgrastim, Bone Marrow Harvest)
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: 10-year Overall Cancer Incidence
Description: The Kaplan-Meier method will be used to estimate overall cancer free probabilities in standard BM and G-BM donors.
Time Frame: Up to 10 years post bone marrow harvest
Population: Data were not collected as no patients were followed to 10 years.
Arm/Group | Arm I (Conventional Bone Marrow Harvest) | Arm II (Filgrastim, Bone Marrow Harvest)
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: 10-year Hematologic Cancer Rate
Description: The Kaplan-Meier method will be used to estimate hematologic cancer probabilities in standard BM and G-BM donors.
Time Frame: Up to 10 years post bone marrow harvest
Population: Data were not collected as no patients were followed to 10 years.
Arm/Group | Arm I (Conventional Bone Marrow Harvest) | Arm II (Filgrastim, Bone Marrow Harvest)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Absolute T Cell Numbers
Description: Median and interquartile range of the outcome measure in standard BM and G-BM donors.
Time Frame: Up to 1 year after donation
Population: Data were not collected for this study.
Arm/Group | Arm I (Conventional Bone Marrow Harvest) | Arm II (Filgrastim, Bone Marrow Harvest)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Th1 vs. Th2 Profile of T Cells
Description: Proportion of donors with Th1-T cell profile in standard BM and G-BM donors.
Time Frame: Up to 1 year after donation
Population: Data were not collected for this study.
Arm/Group | Arm I (Conventional Bone Marrow Harvest) | Arm II (Filgrastim, Bone Marrow Harvest)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Dendritic Cell (DC) Populations
Description: Median and interquartile range of the outcome measure in standard BM and G-BM donors.
Time Frame: Up to 1 year after donation
Population: Data were not collected for this study.
Arm/Group | Arm I (Conventional Bone Marrow Harvest) | Arm II (Filgrastim, Bone Marrow Harvest)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: T Regulatory Cell Content
Description: Median and interquartile range of the outcome measure in standard BM and G-BM donors.
Time Frame: Up to 1 year after donation
Population: Data were not collected for this study.
Arm/Group | Arm I (Conventional Bone Marrow Harvest) | Arm II (Filgrastim, Bone Marrow Harvest)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: First year after Bone Marrow Harvest
Description: Modified Toxicity Criteria and Pain Assessment was used with higher grades corresponding to more severe AEs.
Arm/Group | Arm I (Conventional Bone Marrow Harvest) | Arm II (Filgrastim, Bone Marrow Harvest)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 4/6 | 6/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Conventional Bone Marrow Harvest) (N=6) | Arm II (Filgrastim, Bone Marrow Harvest) (N=7)
Back pain (General disorders) | 1 | 3
Bones (Including Sternum and Ribs) pain (General disorders) | 0 | 1
Dizziness, vertigo, or lightheadedness (General disorders) | 1 | 2
Fatigue (General disorders) | 1 | 6
Fever in the absence of infections (General disorders) | 1 | 1
Headache (General disorders) | 1 | 1
Hip pain (General disorders) | 2 | 2
IV Site pain (General disorders) | 1 | 1
Injection site reaction (General disorders) | 1 | 2
Insomnia (Inability to sleep) (General disorders) | 0 | 1
Joints (Excluding hip) pain (General disorders) | 1 | 1
Limbs (Arm, legs, hands feet) pain (General disorders) | 1 | 1
Loss of Appetite (Anorexia) (General disorders) | 1 | 4
Muscles pain (General disorders) | 0 | 1
Nausea (General disorders) | 0 | 3
Neck pain (General disorders) | 0 | 1
Other pain (General disorders) | 1 | 0
Rashes on skin (General disorders) | 1 | 1
Throat pain (General disorders) | 1 | 4
Vomiting (General disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior approval.